CLINICAL TRIAL: NCT01331252
Title: Can the Incidence of Nosocomial Pneumonia in Severe Tetanus be Reduced by Nursing Patients Semi-recumbent? A Randomised Comparison of Supine or Semi-recumbent Body Position
Brief Title: Pneumonia in Tetanus Study
Acronym: BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BP
Record Dates: First submitted 2011-04-05; First posted 2011-04-08 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Tetanus
MeSH Terms: conditions — Tetanus | interventions — Supine Position

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- supine body position (Experimental): Consecutive patients admitted with severe tetanus to the tetanus intensive care ward will be eligible to be included in the study. An envelope for the next study number will be opened in which patients will be randomly allocated to either semi-recumbent (30 degree) or supine (0 degree) body position
  Interventions: Other: supine
- semi-recumbent (Experimental): Consecutive patients admitted with severe tetanus to the tetanus intensive care ward will be eligible to be included in the study. An envelope for the next study number will be opened in which patients will be randomly allocated to either semi-recumbent (30 degree) or supine (0 degree) body position
  Interventions: Other: semi-recumbent

INTERVENTIONS:
Other: semi-recumbent — Patient rests in a semi-recumbent body position
  Arms: semi-recumbent
Other: supine — Patient rests in a supine position
  Arms: supine body position

SUMMARY:
This is a randomised controlled trial of the incidence of nosocomial pneumonia in patients with severe tetanus admitted to the intensive care ward nursed in a supine or semi-recumbent position.

DETAILED DESCRIPTION:
Background: Hospital-acquired pneumonia remains a common and important cause of morbidity and mortality in patients with severe tetanus who require a tracheostomy whether or not they are mechanically ventilated. We propose to investigate if the incidence of hospital-acquired pneumonia can be reduced by nursing tetanus patients semi-recumbent at 30o rather than supine as is the current practice.

The aim of this study will be to assess the frequency of clinically suspected and microbiologically confirmed hospital acquired pneumonia in patients nursed in a semi-recumbent or supine body position. A secondary end-point will be the mortality in each group. Patients at risk of developing hospital acquired pneumonia (in hospital without developing pneumonia for more than two days) will be evaluated

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients will be entered into the study as they are admitted to the intensive care ward with a clinical diagnosis of tetanus.
2. Informed consent will be obtained from the patient or next-of-kin before randomisation.
3. An envelope for the next study number will be opened in which patients will be randomly allocated to either semi-recumbent (300) or supine (00) body position. The randomisation will be created by a computer generated list.
4. All health care personnel will be instructed not to change the position, unless for medical requirements.
5. The correctness of the position will be checked twice daily.
6. Surveillance for clinical detection of pneumonia or other infection will be done daily. If infection is suspected relevant microbiological samples will be taken.
7. The study period will end 72 hours after the patient has left the intensive care ward, or if there is a permanent change in body position for more than 1 hour or death.

Exclusion Criteria:

1. Recent abdominal surgery (<7 days)
2. Shock refractory to vasoactive drugs or volume therapy
3. Recent intensive care (<30 days)
4. Neonates
5. Pneumonia at the time of admission to intensive care.

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2000-08; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
assess the frequency of clinically suspected and microbiologically confirmed hospital acquired pneumonia | 72 hours
  assess the frequency of clinically suspected and microbiologically confirmed hospital acquired pneumonia in patients nursed in a semi-recumbent or supine body position

SECONDARY OUTCOMES:
mortality between supine or semi-recumbent body position | 72 hours
  mortality in each group. Patients at risk of developing hospital acquired pneumonia (in hospital without developing pneumonia for more than two days) will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Parry, MD, Principal Investigator — Oxford University CLinical Research Unit - Viet Nam

REFERENCES:
- [Derived] Loan HT, Parry J, Nga NT, Yen LM, Binh NT, Thuy TT, Duong NM, Campbell JI, Thwaites L, Farrar JJ, Parry CM. Semi-recumbent body position fails to prevent healthcare-associated pneumonia in Vietnamese patients with severe tetanus. Trans R Soc Trop Med Hyg. 2012 Feb;106(2):90-7. doi: 10.1016/j.trstmh.2011.10.010. Epub 2011 Dec 22. PMID 22197012